CLINICAL TRIAL: NCT07137767
Title: Quantitative Refractive Crosslinking in Presbyopia-Aged Patients: An Open Label, Multi-center, Phase I Study of the TECLens Corneal Crosslinking System for Correction of Refractive Error in Patients of Presbyopia Age
Brief Title: Quantitative Refractive Crosslinking in Presbyopia Aged Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TECLens, Inc. (Industry)
Collaborators: Renato Ambrósio, MD - Rio Vision; Tijuca Rio de Janeiro, Brazil (Unknown); Juan Batlle, Jr. MD - Laser Center; Santo Domingo, Dominican Rep. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEC-007
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Presbyopia
Keywords: Corneal crosslinking; Presbyopia; Myopia; Hyperopia
MeSH Terms: conditions — Presbyopia; Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Epithelium-on Corneal Crosslinking
  Interventions: Device: Quantitative refractive crosslinking

INTERVENTIONS:
Device: Quantitative refractive crosslinking — Non-invasive corneal crosslinking device delivering controlled UV light through a contact lens platform for refractive reshaping of the cornea.

SUMMARY:
An 'on-eye' UV delivery system for corneal crosslinking can be used safely and effectively to help free presbyopic patients from the need for reading glasses.

DETAILED DESCRIPTION:
The clinical trial is evaluating the TECLens CXLens Crosslinking System, an investigational treatment using ultraviolet (UV) light (375 nm) with riboflavin (vitamin B2) to strengthen and reshape the cornea. By creating controlled biomechanical changes, this study aims to test whether the cornea can be reshaped to reduce refractive errors such as mild myopia or hyperopia in patients of presbyopic age.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-65 years
* Healthy cornea
* Refractive error between +4.0 D and -5.0 D
* Phakic or monofocal pseudophakic (≥6 months post IOL placement)
* Visual acuity correctable by ±0.25 D

Exclusion Criteria:

* Corneal dystrophy, scarring, or prior corneal crosslinking
* Astigmatism >1.0 D
* Active ocular infection, inflammation, or uncontrolled dry eye
* Advanced glaucoma or diabetic retinopathy
* History of delayed corneal healing
* Pregnancy, breastfeeding, or planning pregnancy during study period
* Certain medications (e.g., isotretinoin)
* Recent participation in other investigational drug/device studies (within 30 days)
* Patients with uncontrolled dry eye or surface disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Reduce refractive error | 3-months post procedure
  Achieve manifest refraction outcome at 3 months post treatment within 0.75D of the pre-planned targeted refraction, in patients aged 40 to 65 years old

CONTACTS AND LOCATIONS:
Locations (2):
- Rio Vision Hospital Oftalmológico, Rio de Janeiro, Brazil
- Laser Center, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Undecided